CLINICAL TRIAL: NCT03498521
Title: A Phase II, Randomized, Active-Controlled, Multi-Center Study Comparing the Efficacy and Safety of Targeted Therapy or Cancer Immunotherapy Guided by Genomic Profiling Versus Platinum-Based Chemotherapy in Patients With Cancer of Unknown Primary Site Who Have Received Three Cycles of Platinum Doublet Chemotherapy
Brief Title: A Phase II Randomized Study Comparing the Efficacy and Safety of Targeted Therapy or Cancer Immunotherapy Versus Platinum-Based Chemotherapy in Patients With Cancer of Unknown Primary Site
Acronym: CUPISCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MX39795; 2017-003040-20 (EudraCT Number)
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — alectinib; HhAntag691; ipatasertib; olaparib; Erlotinib Hydrochloride; Bevacizumab; Vemurafenib; cobimetinib; pertuzumab; atezolizumab; Carboplatin; Paclitaxel; Cisplatin; Gemcitabine; entrectinib; ivosidenib; pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Molecularly-Guided Therapy (Experimental): Participants will be assigned to molecularly-guided therapy based on genomic profile.
  Interventions: Drug: Alectinib; Drug: Vismodegib; Drug: Ipatasertib; Drug: Olaparib; Drug: Erlotinib; Drug: Bevacizumab; Drug: Vemurafenib; Drug: Cobimetinib; Drug: Trastuzumab Subcutaneous (SC); Drug: Pertuzumab; Drug: Atezolizumab; Drug: Paclitaxel; Drug: Entrectinib; Drug: Ivosidenib; Drug: Pemigatinib
- Platinum-Based Chemotherapy (Active Comparator): Participants will receive platinum-based chemotherapy (Carboplatin or Cisplatin in combination with Gemcitabine or Paclitaxel).
  Interventions: Drug: Trastuzumab Subcutaneous (SC); Drug: Pertuzumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Alectinib — Alectinib will be administered orally at the label-recommended dose (600 mg) twice daily until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months).
  Arms: Molecularly-Guided Therapy
Drug: Vismodegib — Vismodegib will be administered orally at the label-recommended dose (150 mg) once daily until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months).
  Arms: Molecularly-Guided Therapy
Drug: Ipatasertib — Ipatasertib will be administered orally at the label-recommended dose (400 mg) once daily on Days 1-21 of each 28-day Cycle in combination with paclitaxel, and as monotherapy after the final administration of paclitaxel, until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months).
  Arms: Molecularly-Guided Therapy
Drug: Olaparib — Olaparib will be administered orally at the label-recommended dose (400 mg) twice daily until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months).
  Arms: Molecularly-Guided Therapy
Drug: Erlotinib — Erlotinib will be administered orally in combination with Bevacizumab at the label recommended dose (150 mg) once daily until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months)
  Arms: Molecularly-Guided Therapy
Drug: Bevacizumab — Bevacizumab will be administered intravenously at 15mg/kg every 3 weeks in combination with Erlotinib until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months)
  Arms: Molecularly-Guided Therapy
Drug: Vemurafenib — Vemurafenib will be administered orally, 960 mg twice daily, in combination with Cobimetinib, until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months)
  Arms: Molecularly-Guided Therapy
Drug: Cobimetinib — Cobimetinib will be administered orally, 60mg once daily, in combination with Vemurafenib, on Days 1-21 of each 28-day Cycle, until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months)
  Arms: Molecularly-Guided Therapy
Drug: Trastuzumab Subcutaneous (SC) — Trastuzumab will be administered subcutaneously, 600 mg every 3 weeks, in combination with Pertuzumab and chemotherapy, until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months)
Drug: Pertuzumab — Pertuzumab will be initially be administered intravenously, 840 mg, followed by 420 mg every 3 weeks, in combination with Trastuzumab and chemotherapy, until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months)
Drug: Atezolizumab — Atezolizumab will be administered intravenously at the label-recommended dose (1200 mg), alone or in combination with chemotherapy, every 3 weeks until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months).
  Arms: Molecularly-Guided Therapy
Drug: Carboplatin — Carboplatin will be administered intravenously at the area under the curve (AUC) dose once every 3 weeks for up to 9 Cycles (Cycle = 21 days) in some combination with the following: Paclitaxel, Gemcitabine, Atezolizumab, Pertuzumab, and Trastuzumab SC.
  Arms: Platinum-Based Chemotherapy
Drug: Paclitaxel — Paclitaxel will be administered intravenously, 175 mg/m^2, once every 3 weeks for up to 9 cycles (Cycle = 21 days) in some combination with the following: Carboplatin, Ipatasertib, Atezolizumab, Pertuzumab, and Trastuzumab SC
Drug: Cisplatin — Cisplatin will be administered intravenously, 60-75 mg/m^2, once every three weeks, for up to 9 cycles (Cycle = 21 days) in some combination with the following: Gemcitabine, Paclitaxel, Atezolizumab, Pertuzumab, and Trastuzumab SC.
  Arms: Platinum-Based Chemotherapy
Drug: Gemcitabine — Gemcitabine will be administered intravenously, 1000 mg/m^2, twice every three weeks for up to 9 cycles (Cycle = 21 days) in some combination with the following: Cisplatin, Carboplatin, Atezolizumab, Pertuzumab, and Trastuzumab SC.
  Arms: Platinum-Based Chemotherapy
Drug: Entrectinib — Entrectinib will be administered orally at the label-recommended dose (600 mg) once daily until loss of clinical benefit or unacceptable toxicity, through the end of the study (approximately 70 months).
  Arms: Molecularly-Guided Therapy
Drug: Ivosidenib — Ivosidenib will be administered orally at the label-recommended dose (500mg) once daily across a 28-day treatment cycle until loss of clinical benefit or unacceptable toxicity.
  Arms: Molecularly-Guided Therapy
Drug: Pemigatinib — Pemigatinib will be administered orally at the label-recommended dose (13.5mg) once daily across a 21-day treatment cycle until loss of clinical benefit or unacceptable toxicity.
  Arms: Molecularly-Guided Therapy

SUMMARY:
This study will compare the efficacy and safety of molecularly-guided therapy versus standard platinum-containing chemotherapy in participants with poor-prognosis cancer of unknown primary site (CUP; non-specific subset) who have achieved disease control after 3 cycles of first-line platinum based induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed unresectable cancer of unknown primary site (CUP) diagnosed according to criteria defined in the 2015 European Society for Medical Oncology (ESMO) Clinical Practice Guidelines for CUP
* No prior lines of systemic therapy for the treatment of CUP
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Candidate for platinum-based chemotherapy (according to the reference information for the intended chemotherapy)
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
* Formalin-Fixed Paraffin-Embedded (FFPE) tumor tissue sample </= 4 months old that is expected to be sufficient for generation of a comprehensive genomic profile at a central reference pathology laboratory

Exclusion Criteria:

* Squamous cell CUP
* Participants who can be assigned to a specific subset of CUP for which a specific treatment is recommended by the 2015 ESMO Clinical Practice Guidelines for CUP or with a clinical and IHC profile indicative of a specific primary tumor (favorable prognosis CUP subsets): Poorly differentiated carcinoma with midline distribution; women with papillary adenocarcinoma of the peritoneal cavity; women with adenocarcinoma involving only the axillary lymph nodes; squamous cell carcinoma of the cervical lymph nodes; poorly differentiated neuroendocrine tumors; men with blastic bone metastases and elevated prostate-specific antigen (PSA); participants with a single, small, potentially resectable tumor; colon cancer-type CUP, including participants with a CK7 negative, CK20 positive, CDX-2 positive immunohistochemistry profile; CK7-positive, CK20-negative and TTF-1 positive tumors in a context suggestive of lung adenocarcinoma or thyroid cancer; IHC profile definitely indicative of breast cancer OR an IHC profile indicative of breast cancer and either a history of breast cancer or lymph nodes in the drainage areas of the breast; high-grade serious carcinoma histology and elevated CA125 tumor marker and/or a mass in the gynecological tract or any tumor mass or lymph node in the abdominal cavity; IHC profile suggestive of renal cell carcinoma and renal lesions, with a Bosniak classification higher than IIF; IHC profile compatible with cholangiocarcinoma or pancreatobiliary (or upper gastrointestinal carcinoma) AND 1 or 2 liver lesions without extrahepatic disease or with only pulmonary metastases and/or lymph nodes in the drainage areas of the liver
* Known presence of brain or spinal cord metastasis (including metastases that have been irradiated only)
* Histology and immunohistology profiles (per 2015 ESMO guidelines) that are not adenocarcinoma or poorly differentiated carcinoma/adenocarcinoma
* History or known presence of leptomeningeal disease
* Known human immunodeficiency virus (HIV) infection
* Significant cardiovascular disease
* Prior allogeneic stem cell or solid organ transplantation
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or for up to 7 months after the final dose of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (125):
- Australia (3):
  - Blacktown Hospital, Blacktown, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
- Austria (3):
  - Lkh-Univ. Klinikum Graz, Graz
  - Lkh Salzburg - Univ. Klinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Brazil (5):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
- Bulgaria (2):
  - MHAT Nadezhda, Sofia
  - MBAL Serdika EOOD, Sofia
- Chile (2):
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - James Lind Centro de Investigación Del Cáncer, Temuco
- Colombia (3):
  - Clinica del Country, Bogotá
  - Inst. Nacional de Cancerologia, Bogotá
  - Oncomedica S.A., Montería
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice, Prague
- Aarhus Universitetshospital, Aarhus N, Denmark
- North Estonia Medical Centre, Oncology and hematology Clinic, Tallinn, Estonia
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (15):
  - Ico - Paul Papin, Angers
  - CHRU Besançon, Besançon
  - Institut Bergonie, Bordeaux
  - CRLCC-Francois Baclesse, Caen
  - Centre Jean Perrin Centre Regional de Lutte Contre Le Cancer D auvergne, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - CHU Lyon - Centre Hospitalier Lyon Sud, Pierre-Benite (Lyon)
  - Centre Eugene Marquis, Rennes
  - CHU Strasbourg Hpital Hautepierre, Strasbourg
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité-Universitätsm. Berlin, Berlin
  - Onkologisches Zentrum - Onkologie Dachau, Dachau
  - Universitätsklinikum Frankfurt, UCT, Frankfurt
  - SLK-Kliniken Heilbronn GmbH;Klinik für Innere Medizin III, Heilbronn
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena
  - Klinikum Mannheim III. Medizinische Klinik, Mannheim
  - Klinikum der LMU München, Campus Großhadern, Krebszentrum München, München
  - Universitätsklinikum Münster, Medizinische Klinik A, Translationale Onkologie, Münster
  - RED-Oncology GmbH, Oldenburg / Holstein
- Greece (5):
  - Anticancer Hospital Ag Savas, Athens
  - IASO General Hospital of Athens, Athens
  - Univ General Hosp Heraklion, Heraklion
  - Uni Hospital of Ioannina, Ioannina
  - Theagenio Anticancer Hospital, Thessaloniki
- Hungary (3):
  - Orszagos Onkologiai Intezet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Bács-Kiskun Vármegyei Oktatókórház, Kecskemét
- Ireland (2):
  - St Vincent'S Uni Hospital, Dublin
  - Waterford Regional Hospital, Waterford
- Israel (3):
  - Rabin MC, Petah Tikva
  - Chaim Sheba medical center, Oncology division, Ramat Gan
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
- Italy (7):
  - U. O. Oncologia Medica, Ospedale Santa Chiara, Pisa, Basilicate
  - Policlinico Univ. - A.O. Mater Domini, Catanzaro, Calabria
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Japan (3):
  - Aichi Cancer Center, Aichi
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
- Riga East Clinical University Hospital Latvian Oncology Centre, Riga, Latvia
- Mexico (2):
  - Health Pharma Professional Research, CD Mexico, Mexico CITY (federal District)
  - AVIX Investigación Clínica S.C, Monterrey, Nuevo León
- Netherlands (3):
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Ziekenhuis VieCuri Medisch Centrum, Venlo
- Norway (3):
  - Sørlandet Sykehus Kristiansand, Kristiansand
  - Akershus universitetssykehus HF, Lørenskog
  - Oslo universitetssykehus HF, Ullevål, Kreftsenteret, Oslo
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Oncosalud Sac, Lima
- Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow, Poland
- IPO do Porto, Porto, Portugal
- Romania (4):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj Napoca, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Oncocenter Timisoara, Timi?oara
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (10):
  - Hospital Sant Joan Despi- Moises Broggi, Sant Joan Despí, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Complexo Hospitalario de Vigo. Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Clínic i Provincial, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (2):
  - Universitaetsspital Basel, Basel
  - UniversitätsSpital Zürich, Zurich
- Thailand (2):
  - Ramathibodi Hospital;Medicine/Oncology, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
- Turkey (Türkiye) (8):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Ankara University Medical Faculty, Ankara
  - Ankara Oncology Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Istanbul University Cerrahpa?a-Cerrahpa?a Medical Faculty, Istanbul
  - ?zmir Medical Point, Kar?iyaka
  - Hacettepe Uni Medical Faculty Hospital, S?hhiye, Ankara
- United Kingdom (8):
  - Royal United Hospital, Bath
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Hammersmith Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Southampton General Hospital, Southampton
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Kramer A, Bochtler T, Pauli C, Shiu KK, Cook N, de Menezes JJ, Pazo-Cid RA, Losa F, Robbrecht DG, Tomasek J, Arslan C, Ozguroglu M, Stahl M, Bigot F, Kim SY, Naito Y, Italiano A, Chalabi N, Duran-Pacheco G, Michaud C, Scarato J, Thomas M, Ross JS, Moch H, Mileshkin L. Molecularly guided therapy versus chemotherapy after disease control in unfavourable cancer of unknown primary (CUPISCO): an open-label, randomised, phase 2 study. Lancet. 2024 Aug 10;404(10452):527-539. doi: 10.1016/S0140-6736(24)00814-6. Epub 2024 Jul 31. PMID 39096924

RESULTS

PARTICIPANT FLOW:
Groups:
- Molecularly-Guided Therapy (MGT) Category 1: Category 1 included participants with cancer of unknown primary site (CUP) with a complete response (CR), partial response (PR), or stable disease (SD) after 3 cycles of platinum induction chemotherapy (provided at the beginning of the study). MGT was chosen based on each participant's comprehensive genomic profile and administered until loss of clinical benefit, unacceptable toxicity, participant or investigator decision to discontinue, or death, whichever occurred first.
- Chemotherapy Category 1: Category 1 included participants with cancer of unknown primary site (CUP) with a complete response (CR), partial response (PR), or stable disease (SD) after 3 cycles of platinum induction chemotherapy (provided at the beginning of the study).
  Participants in this arm continued to receive the same chemotherapy regimen used during induction for a minimum of 3 additional cycles.
- Category 2: Category 2 included participants with progressive disease (PD) after 3 cycles of platinum induction chemotherapy. Participants in this arm received either MGT based on their comprehensive genomic profile until loss of clinical benefit, unacceptable toxicity, participant or investigator decision to discontinue, or death, whichever occurred first, or the same chemotherapy regimen used during induction for a minimum of 3 additional cycles.
Period: Overall Study
Arm/Group | Molecularly-Guided Therapy (MGT) Category 1 | Chemotherapy Category 1 | Category 2
Started | 326 | 110 | 93
Completed | 0 | 0 | 0
Not Completed | 326 | 110 | 93
Not completed — Death | 227 | 79 | 84
Not completed — Exclusion criteria | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — No profile due to technical failure | 1 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 6 | 2
Not completed — Study terminated by sponsor | 79 | 21 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Molecularly-Guided Therapy (MGT) Category 1 | Chemotherapy Category 1 | Category 2 | Total
Number analyzed (Participants) | 326 | 110 | 93 | 529
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (11.5) | 61.1 (11.3) | 59.2 (12.7) | 60.42 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 53 | 44 | 258
  Male | 165 | 57 | 49 | 271
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 1 | 8
  Asian | 31 | 12 | 7 | 50
  Black or African American | 5 | 0 | 0 | 5
  Unknown | 43 | 14 | 15 | 72
  White | 242 | 81 | 70 | 393
  Missing | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 9 | 4 | 35
  Not Hispanic or Latino | 252 | 85 | 76 | 413
  Not Stated | 31 | 11 | 7 | 49
  Unknown | 21 | 5 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by the Investigator According to Response Evaluation Criteria In Solid Tumors v1.1 (RECIST v1.1)
Description: This efficacy objective was to evaluate the efficacy of MGT vs platinum chemotherapy in term of PFS in participants with CUP whose best response to 3 cycles of platinum induction chemotherapy was assessed CR, PR, or SD.
Time Frame: From randomization to the first occurrence of disease progression or death from any cause, until 330 PFS events were observed (approx. 4.3 years for MGT Cat 1 and 3.4 years for Chemotherapy Cat 1).
Population: The intent-to-treat (ITT) population included all Category 1 randomized participants, whether or not the assigned study treatment was received. Endpoints for Category 2 were exploratory and were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Molecularly-Guided Therapy (MGT) Category 1 | Chemotherapy Category 1
Number analyzed (Participants) | 326 | 110
Months | 6.14 [4.70 to 6.47] | 4.40 [4.17 to 6.37]
Statistical Analysis 1: Comparison: Molecularly-Guided Therapy (MGT) Category 1 vs Chemotherapy Category 1; Test type: Superiority; p = 0.0177, Stratified log-rank; Stratified Cox proportional hazard = 0.75, 95% CI 2-sided [0.59 to 0.95]

2. Secondary Outcome: Overall Survival (OS)
Time Frame: From randomization to death from any cause (approx. 4 years)
Population: The ITT population included all Category 1 randomized participants, whether or not the assigned study treatment was received. Endpoints for Category 2 were exploratory and were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Molecularly-Guided Therapy MGT) Category 1: Category 1 included participants with cancer of unknown primary site (CUP) with a complete response (CR), partial response (PR), or stable disease (SD) after 3 cycles of platinum induction chemotherapy (provided at the beginning of the study). MGT was chosen based on each participant's comprehensive genomic profile and administered until loss of clinical benefit, unacceptable toxicity, participant or investigator decision to discontinue, or death, whichever occurred first.
Arm/Group | Molecularly-Guided Therapy MGT) Category 1 | Chemotherapy Category 1
Number analyzed (Participants) | 326 | 110
Months | 15.18 [13.90 to 18.43] | 12.78 [9.86 to 15.38]

3. Secondary Outcome: Objective Response Rate (ORR)
Time Frame: Two consecutive occurrences of complete or partial response >/=4 weeks apart (up to approximately 4 months)
Population: The ITT population included all Cat. 1 randomized participants, whether or not the assigned study treatment was received. Cat. 2 endpoints were exploratory and not analyzed.
  NA: Participants had no lesions to report at baseline NE: Post-baseline assessments reported not evaluable for any reason or if SD assessment was within 6 weeks of baseline Missing: No post-baseline assessments available
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Molecularly-Guided Therapy MGT) Category 1 | Chemotherapy Category 1
Number analyzed (Participants) | 326 | 110
Percentage of participants
  Complete response (CR) | 4.9 [2.83 to 7.85] | 3.6 [1.00 to 9.05]
  Partial response (PR) | 12.9 [9.45 to 17.01] | 4.5 [1.49 to 10.29]
  Stable disease (SD) | 44.5 [39.00 to 50.06] | 49.1 [39.43 to 58.80]
  Non-CR/Non-PD | 7.1 [4.52 to 10.40] | 6.4 [2.60 to 12.67]
  Not Applicable (NA) | 2.5 [1.07 to 4.78] | 2.7 [0.57 to 7.76]
  Progressive disease (PD) | 17.8 [13.80 to 22.38] | 21.8 [14.51 to 30.70]
  Not evaluable participants | 0.6 [0.07 to 2.20] | 0 [0.00 to 3.30]
  Missing participants | 9.8 [6.81 to 13.57] | 11.8 [6.45 to 19.36]

4. Secondary Outcome: Duration of Response (DOR)
Time Frame: From the first documentation of a complete response (CR) or partial response (PR) to disease progression or death from any cause, whichever occurs first (up to approximately 4 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Molecularly-Guided Therapy MGT) Category 1 | Chemotherapy Category 1
Number analyzed (Participants) | 58 | 9
Months | 16.39 [8.08 to NA] — Value is NA due to insufficient no. of participants with the event. | NA [4.14 to NA] — Value is NA due to insufficient no. of participants with the event.

5. Secondary Outcome: Disease Control Rate (DCR)
Time Frame: From randomization to death from any cause, through the end of study (approximately 4 years)
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Molecularly-Guided Therapy MGT) Category 1 | Chemotherapy Category 1
Number analyzed (Participants) | 326 | 110
Percentage of responders | 64.7 [59.27 to 69.91] | 60.0 [50.22 to 69.22]

ADVERSE EVENTS:
Time Frame: Approximately 4.5 years
Description: The all-cause mortality table contains all participants.
  The safety evaluable (SE) population (used to report serious and other AE) included all participants who received at least one dose of any component of study drug.
Arm/Group | Molecularly-Guided Therapy (MGT) Category 1 | Chemotherapy Category 1 | Category 2
All-Cause Mortality (participants affected / at risk) | 227/326 | 79/110 | 84/93
Serious Adverse Events (participants affected / at risk) | 119/312 | 15/102 | 39/93
Other Adverse Events (participants affected / at risk) | 279/312 | 81/102 | 73/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molecularly-Guided Therapy (MGT) Category 1 (N=312) | Chemotherapy Category 1 (N=102) | Category 2 (N=93)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 7 (7) | 1 (1) | 2 (2)
Peritonitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (6) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4)
Infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Endocarditis noninfective (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mononeuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vestibular migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molecularly-Guided Therapy (MGT) Category 1 (N=312) | Chemotherapy Category 1 (N=102) | Category 2 (N=93)
Anaemia (Blood and lymphatic system disorders) | 111 (180) | 30 (37) | 37 (55)
Leukopenia (Blood and lymphatic system disorders) | 16 (26) | 9 (15) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 62 (100) | 24 (41) | 11 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 49 (80) | 14 (25) | 13 (20)
Abdominal pain (Gastrointestinal disorders) | 35 (40) | 3 (3) | 10 (11)
Constipation (Gastrointestinal disorders) | 43 (55) | 12 (13) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 76 (118) | 6 (8) | 9 (11)
Nausea (Gastrointestinal disorders) | 88 (127) | 20 (34) | 23 (36)
Vomiting (Gastrointestinal disorders) | 41 (58) | 13 (17) | 10 (12)
Asthenia (General disorders) | 60 (86) | 15 (19) | 15 (17)
Fatigue (General disorders) | 69 (106) | 14 (19) | 22 (28)
Oedema peripheral (General disorders) | 26 (31) | 3 (6) | 8 (8)
Pyrexia (General disorders) | 29 (46) | 4 (6) | 10 (10)
COVID-19 (Infections and infestations) | 27 (28) | 2 (2) | 5 (5)
Neutrophil count decreased (Investigations) | 33 (59) | 9 (13) | 9 (22)
Platelet count decreased (Investigations) | 38 (78) | 9 (18) | 11 (15)
Weight decreased (Investigations) | 20 (20) | 3 (3) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 60 (74) | 10 (12) | 14 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 (37) | 5 (7) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (34) | 2 (3) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 (67) | 6 (6) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 4 (4) | 5 (6)
Insomnia (Psychiatric disorders) | 17 (21) | 1 (1) | 5 (5)
Hypothyroidism (Endocrine disorders) | 20 (20) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 19 (21) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (36) | 5 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 17 (26) | 7 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (23) | 6 (6) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 17 (20) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 16 (18) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (29) | 7 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (35) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 17 (21) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 19 (21) | 3 (5) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 39 (46) | 15 (18) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (25) | 7 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (42) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (24) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 28 (43) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 35 (48) | 2 (5) | 0 (0)
Hypertension (Vascular disorders) | 22 (28) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 6 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT03498521/Prot_SAP_001.pdf